CLINICAL TRIAL: NCT03215966
Title: Single-center, Open-label, Single-dose, Two-period, Randomized, Crossover, Phase I Study to Demonstrate Bioequivalence Between a Fixed Dose Combination Product Formulation of Macitentan/Tadalafil (10 mg/40 mg) and the Free Combination of 10 mg Macitentan (Opsumit®) and 40 mg Tadalafil (Adcirca®) in Healthy Male and Female Subjects
Brief Title: A Study to Compare the Macitentan-tadalafil Fixed Dose Combination Tablet Relative to the Concomitant Administration of the Reference Tablets of Macitentan and Tadalafil in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-077-103
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects
Keywords: bioequivalence
MeSH Terms: interventions — macitentan; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A/B (Experimental): Subjects receive one tablet of macitentan / tadalafil FDC (fixed dose combination) during Period 1, then after a washout period of at least 7 days they receive one tablet of macitentan (Opsumit®) and two tablets of tadalafil (Adcirca®) during Period 2
  Interventions: Combination Product: Macitentan / tadalafil FDC; Drug: Macitentan (Opsumit®); Drug: Tadalafil (Adcirca®)
- Sequence B/A (Experimental): Subjects receive one tablet of macitentan (Opsumit®) and two tablets of tadalafil (Adcirca®) during Period 1, then after a washout period of at least 7 days, they receive one tablet of macitentan / tadalafil FDC (fixed dose combination) during Period 2
  Interventions: Combination Product: Macitentan / tadalafil FDC; Drug: Macitentan (Opsumit®); Drug: Tadalafil (Adcirca®)

INTERVENTIONS:
Combination Product: Macitentan / tadalafil FDC — Tablets for oral administration containing 10 mg of macitentan and 40 mg of tadalafil
Drug: Macitentan (Opsumit®) — Film-coated tablets for oral administration formulated at a strength of 10 mg
  Other Names: ACT-064992
Drug: Tadalafil (Adcirca®) — Film-coated tablets for oral administration formulated at a strength of 20 mg

SUMMARY:
The primary objective of this study is to demonstrate that macitentan and tadalafil administered as a fixed combination is bioequivalent to both compounds given as separate tablets given at the same doses as in the fixed combination (i.e. whether the amounts of macitentan and tadalfil which reach the blood are comparable).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent
* Male and female subjects aged between 18 and 55 years (inclusive) at screening
* Healthy on the basis of the physical examination, vital signs, 12-lead ECG, and laboratory tests performed at screening
* Women must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day-1 or must be of non-childbearing potential.
* Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) at screening
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 bpm (inclusive)

Key Exclusion Criteria:

* Known hypersensitivity to any active substance or drugs of the same class, or any excipients of the drug formulation(s)
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study treatment(s)
* Values of hepatic aminotransferase (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST]) > 3 X upper limit of normal at screening
* Loss of vision in one eye because of non-arteritic anterior ischemic optic neuropathy
* Known hereditary degenerative retinal disorders, including retinitis pigmentosa
* Priapism and anatomical deformation of the penis
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions
* Treatment with another investigational drug within 3 months prior to screening or participation in more than 4 investigational drug studies within 1 year prior to screening
* Excessive caffeine consumption, defined as > or = 800 mg per day at screening.
* Nicotine intake (e.g., smoking, nicotine patch, nicotine chewing gum, or electronic cigarettes) within 3 months prior to screening and inability to refrain from nicotine intake from screening until end-of-study (EOS; washout period included)
* Previous treatment with any prescribed medications (including vaccines) or over the counter (OTC) medications within 3 weeks prior to first study treatment administration.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-09-24 (Actual); Study Completion 2017-09-24 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of macitentan and tadalafil | Blood samples for pharmacokinetic evaluations are collected at selected time points from Baseline (pre-dose) to 216 hours post-dose of each study period
  The measured individual plasma concentrations of macitentan and tadalafil are used to directly obtain Cmax
Area under the plasma concentration-time curve from 0 to time t [AUC(0-t)] of macitentan and tadalafil | Blood samples for pharmacokinetic evaluations are collected at selected time points from Baseline (pre-dose) to 216 hours post-dose of each study period
  AUC(0-t) is the area calculated from the concentration-time profile of macitentan and tadalafil, from time 0 to to time t of the last measured concentration above the limit of quantification
Area under the plasma concentration-time curve to infinitiy [AUC(0-inf)] of macitentan and tadalafil | Blood samples for pharmacokinetic evaluations are collected at selected time points from Baseline (pre-dose) to 216 hours post-dose of each study period
  AUC(0-inf) is the area calculated from the concentration-time profile of macitentan and tadalafil, from time 0 to extrapolated infinite time

SECONDARY OUTCOMES:
maximal plasma concentration (Cmax) of ACT-132577 | Blood samples for pharmacokinetic evaluations are collected at selected time points from Baseline (pre-dose) to 216 hours post-dose of each study period
  Cmax of the active metabolite of macitentan, ACT-132577, is measured directly from the plasma concentrations of ACT-132577
Area under the plasma concentration-time curve from 0 to time t [AUC(0-t)] of ACT-132577 | Blood samples for pharmacokinetic evaluations are collected at selected time points from Baseline (pre-dose) to 216 hours post-dose of each study period
  AUC(0-t) of the active metabolite of macitentan, ACT-132577, is calculated from the concentration-time profile of ACT-132577 from time 0 to time t of the last measured concentration above the limit of quantification
Area under the plasma concentration-time curve to infinity [AUC(0-inf)] of ACT-132577 | Blood samples for pharmacokinetic evaluations are collected at selected time points from Baseline (pre-dose) to 216 hours post-dose of each study period
  AUC(0-inf) of the active metabolite of macitentan, ACT-132577, is calculated from the concentration-time profile of ACT-132577 from time 0 to extrapolated infinite time

CONTACTS AND LOCATIONS:
Overall Officials: JP Jones, Study Director — Actelion
Locations (1):
- CRS Clinical Research Services Mannheim, Mannheim, Germany